CLINICAL TRIAL: NCT03165747
Title: Effect of VSL#3 on Bone Mineral Density in Postmenopausal Women: a Pilot Randomized, Placebo-Controlled Trial
Brief Title: Effect of VSL#3 on Bone Mineral Density in Postmenopausal Women
Acronym: ProBoneVSL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator terminated trial pursuant to research contract rights.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Roberto Pacifici, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00095798
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Menopausal Osteoporosis
Keywords: Probiotics; Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the Emory Investigational Drug Service (IDS) pharmacy will know which dose of probiotic was given to the subject. The study team, parents, subjects, individuals entering the data, statistician, individuals performing laboratory tests and DEXA scans, research center nurses and investigators will remain blinded as to which treatment the subjects received. Each subject will be assigned a unique identifier, which will be used in the database. In addition, all lab specimens will only include the patient's unique identifier. Permuted block sizes will not be disclosed to the blinded study personnel to minimize the likelihood of their being able to predict the next randomization assignment in the series. Investigators and all study personnel will remain blinded until the final subject has completed her final visit and primary and secondary endpoints have been analyzed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VSL#3 (Experimental): VSL#3 two active sachets [containing 450x109 colony-forming units (CFU)/sachet], taken daily in a single administration.
  Interventions: Drug: VSL#3
- Control (Placebo Comparator): Placebo, no supplemental probiotics.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VSL#3 — 8 strains of live bacteria: Bifidobacterium breve, B. longum, B. infantis, L. acidophilus, L. plantarum, L. paracasei, L. bulgaricus and Streptococcus thermophilus. 900 billion CFU taken orally daily in a single administration.
  Arms: VSL#3
Other: Placebo — Two placebo sachets taken orally daily in a single administration.
  Arms: Control

SUMMARY:
Osteoporosis has a devastating impact on quality of life of postmenopausal women, and is a significant cause of disability and morbidity. Many drugs are approved for the prevention and treatment of osteoporosis, but are associated with high costs and side effects. Some data from animal studies suggests that supplementation with probiotics can safely treat and prevent osteoporosis. The probiotic VSL#3 is commercially available, is safe for human consumption, and has been widely used in human clinical trials, and has known health-promoting effects in both children and adults.

The double-blind, randomized, placebo-controlled trial of VSL#3 will be conducted for 12 months in 40 postmenopausal women to determine if VSL#3 improves bone mineral density and related bone markers. Study visits will include all or some of the following procedures: a medical exam, urine collection, height and weight measurement, a blood draw to assess bone biomarkers, a DEXA (dual energy X-ray absorptiometry) scan to measure bone density, and health questionnaires.

This is one of the first clinical trials proposed to investigate the effects of probiotics in bone in humans. If successful, this proposal will provide the first evidence that nutritional supplementation with the probiotic VSL#3 is a safe and effective strategy for preventing postmenopausal bone loss.

DETAILED DESCRIPTION:
Osteoporosis has a devastating impact on quality of life of postmenopausal women, and is a significant cause of disability and morbidity. Many drugs are approved for the prevention and treatment of osteoporosis, but are associated with high costs and side effects. Some data from animal studies suggests that supplementation with probiotics can safely treat and prevent osteoporosis. The probiotic VSL#3 is commercially available, is safe for human consumption, and has been widely used in human clinical trials, and has known health-promoting effects in both children and adults.

The double-blind, randomized, placebo-controlled trial of VSL#3 will be conducted in a population of ambulatory, otherwise healthy, postmenopausal women for 12 months. Control and VSL#3-treated postmenopausal women will be matched by age (± 3 years). Study visits will include all or some of the following procedures: a medical exam, urine collection, height and weight measurement, a blood draw to assess bone biomarkers, a dual energy X-ray absorptiometry (DEXA) scan to measure bone density, and health questionnaires.

The primary endpoint is the change in bone mineral density (BMD) at the L1-4 lumbar spine over one year of study. Changes in BMD at the femoral neck and total hip area will be secondary endpoints. All BMD data will also be used as a tool for future studies power calculation and design. Additional endpoints will include changes in bone turnover markers and inflammatory/osteoclastogenic cytokines. Measurements of indices of bone turnover and cytokine levels will provide much needed mechanistic information.The data will allow to establish whether VSL#3 prevents bone loss and/or increases bone mass by regulating bone resorption, formation, or both.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study
2. Age range 50-65 years
3. Menopausal status (defined by >1 yr since last menstrual period or follicle stimulating hormone (FSH) level in the postmenopausal range)
4. Ambulatory
5. Body mass Index (BMI) must be ≥ 18 and ≤ 32 kg/m2 at screening
6. Bone mineral density (BMD), expressed as T-scores, must be > - 2.5 in the lumbar spine (L1-L4), the femoral neck, and the total hip, as measured by DEXA
7. Commitment not to use any products that may influence the study outcome
8. Ability to understand and comply with the requirements of the study

Exclusion Criteria:

1. Premenopausal status
2. History of >1 previous atraumatic bone fractures after age 50
3. Presence of established osteoporosis (T-score ≤ - 2.5, in the lumbar spine, femoral neck or total hip as measured by screening DEXA)
4. History of immunological or bone-related disorders including: HIV infection, Type I diabetes mellitus, bone marrow or organ transplantation; Inflammatory bowel disease (ulcerative colitis, Crohn's disease); multiple myeloma; osteomalacia; osteosarcoma; Paget's disease; rheumatoid arthritis; systemic lupus erythematous; parathyroid disorders
5. Uncontrolled type II diabetes mellitus (HgbA1c ≥ 7% within the last 12 months)
6. History of bariatric surgery or other forms of malabsorption (including documented celiac disease, or chronic diarrhea)
7. Alcohol abuse
8. Clinically significant chronic kidney disease (stage ≥ 2, with total serum creatinine level > 2.5 mg/dL and calculated glomerular filtration rate (GFR) < 60 mL/min by the Modification of Diet in Renal Disease (MDRD equation)
9. Clinically significant cardiovascular disease (myocardial infarction, cerebral vascular accident or acute congestive heart failure within the previous 12 months
10. Any malignancies, other than localized skin squamous cell carcinoma, diagnosed within the previous 5 years, or any history of metastatic cancer
11. History of use of oral supplement products containing probiotic bacteria (more than once per week) within four weeks prior to baseline
12. Current use (within the past 8 weeks) of any medication with known influences on the immune or skeletal system (e.g. immune modulation therapy, systemic glucocorticoids, systemic steroid hormones
13. Use of oral or injectable bisphosphonates for more than 1 year within the last 5 years
14. Current or past use (within 1 year) of Denosumab, Teriparatide, Raloxifene, hormone replacement therapy (HRT), calcitonin, or any other anti-resorptive agent other than bisphosphonates used for the prevention and treatment of osteoporosis
15. Use of antibiotics during the previous two months or frequent user of antibiotics (>2 courses during the previous 12 months) for any cause
16. Smoking or use of nicotine-containing products during the last six months
17. Known hypersensitivity to any of the ingredients in the VSL#3 or the placebo study drug
18. serum or plasma 25-hydroxyvitamin D [25(OH)D] concentration < 12 ng/mL
19. uncontrolled thyroid disease (abnormal blood thyroid stimulating hormone (TSH) level within the last 12 months and/or changing dose of thyroid replacement therapy within the last 12 months)

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 35 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pacifici, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Clinical Research Network, Emory Clinic, Emory St. Joseph's Hospital, Emory University Hospital (non-CRN), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Emory University Hospital in Atlanta, Georgia, USA. Enrollment began on October 1, 2017 and all study activity stopped on March 23, 2019.
Pre-assignment Details: 35 individuals consented to participate. The investigational product became the subject of a court judgment upholding false advertising claims concerning the product's similarity to earlier products sold under the same name. Because of questions raised by this ruling, no participants are considered as being assigned to a protocol-defined study arm.
Groups:
- VSL#3: Participants randomized to receive two sachets of the VSL#3 probiotic, taken orally daily in a single administration.
- Placebo: Participants randomized to receive two placebo sachets, taken orally daily in a single administration.
Period: Overall Study
Arm/Group | VSL#3 | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The investigational product became the subject of a court judgment upholding false advertising claims concerning the product's similarity to earlier products sold under the same name. Because of questions raised by this ruling, no participants are considered as being assigned to a protocol-defined study arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | VSL#3 | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (BMD) of the Lumbar Spine (L1-L4 Segment) as Measured by Dual Energy X-ray Absorptiometry (DEXA)
Description: All DEXA scans will be performed on the same device using a GE Lunar iDEXA machine. Participants will be asked to lie still on a scanning table with their arms at their sides for approximately 10 minutes.
Time Frame: Baseline and 12-month visit.
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Bone Density of the Non-dominant Hip (Femoral Neck and Total Hip Area) as Measured by DEXA (Dual Energy X-ray Absorptiometry).
Description: as for outcome 1
Time Frame: Baseline and 12-month visit.
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Serum Collagen Type 1 Cross-linked C-telopeptide (CTX) Concentrations (a Marker of Bone Resorption).
Description: Up to approximately 50 mL of fasted blood will be collected at every visit from a peripheral vein.
Time Frame: Baseline, 6-month, 12-month visits
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Serum Procollagen Type I N Propeptide (PINP) - a Marker of Bone Formation - Concentrations.
Description: Up to approximately 50 mL of fasted blood will be collected at every visit from a peripheral vein.
Time Frame: Baseline, 6-month, 12-month visits
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Serum Free Receptor Activator of Nuclear Factor Kappa-B Ligand (RANKL) Concentrations.
Description: Up to approximately 50 mL of fasted blood will be collected at every visit from a peripheral vein.
Time Frame: Baseline, 6-month, 12-month visits
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Serum Osteoprotegrin (OPG) Concentrations.
Description: Up to approximately 50 mL of fasted blood will be collected at every visit from a peripheral vein.
Time Frame: Baseline, 6-month, 12-month visits
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Serum Tumor Necrosis Factor (TNF)
Description: Up to approximately 50 mL of fasted blood will be collected at every visit from a peripheral vein.
Time Frame: Baseline, 6-month, 12-month visits
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Serum Interleukin-17 (IL-17) Concentrations.
Description: Up to approximately 50 mL of fasted blood will be collected at every visit from a peripheral vein.
Time Frame: Baseline, 6-month, 12-month visits
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Unused Study Drug Sachets.
Description: This will be determined by contacts (twice monthly telephone or at research center visits) of the study coordinator with each subject and responses to three standardized question areas: 1) "Are you having any difficulty, problems or new symptoms with the study medication?" 2) If yes, "What has the problem been?" and 3) "Have you missed any of your study drug doses, and if so how many in the previous 2 week period?" Appropriate notations based on subject responses will be documented in the case report form (CRF). Subjects will be instructed at study entry and reminded via serial contacts to return all of their used and unused drug sachets at each research center visit. Unused and used study drug sachets will be tallied and recorded in the CRF by the study coordinator serially for the entire study.
Time Frame: Every two weeks during the study 12-months
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Gastrointestinal Symptom Rating
Description: Study drug tolerance will be assessed by obtaining serial measures of the Gastrointestinal Symptom Rating Scale (GSRS). These will be obtained with in-person interviews at the baseline and month 6 and 12 visits and by telephone contact with all subjects by the study coordinator every 2 weeks. Data will be analyzed within the 5 symptom domains depicting symptoms related to gastric reflux, abdominal pain, indigestion, diarrhea, and constipation.The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms. A GSRS total score, the sum of all 5 domains, will also be assessed.
Time Frame: Every two weeks during the study 12-months
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Study Retention Rate.
Description: The number of participants who complete all study visits, phone calls, and maintain drug compliance. Retention will be documented via conventional Consolidated Standards of Reporting Trials (CONSORT) criteria and documentation of missed study visits, missed telephone communications and compliance with study drug administration. All data will be maintained in the CRFs.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Upon beginning to take the study products, participants were called every other week to monitor for any adverse effects. In addition to twice monthly phone calls, participants were asked to complete Subject Diary Cards to capture adverse events during the course of the trial and up to 1 month following the cessation of the study drug (up to Month 13).
Description: The investigational product became the subject of a court judgment upholding false advertising claims concerning the product's similarity to earlier products sold under the same name. Because of questions raised by this ruling, no participants are considered as being assigned to a protocol-defined study arm.
Arm/Group | VSL#3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT03165747/Prot_SAP_000.pdf